CLINICAL TRIAL: NCT04217928
Title: Comparison of Arthroscopic Debridement and Arthroscopic Hemi-Trapeziectomy With Mini TightRope on Patients With Thumb Carpometacarpal Joint Osteoarthritis - A Prospective Randomized Single-Blinded Controlled Trial
Brief Title: Arthroscopic Debridement vs Arthroscopic Hemi-Trapeziectomy on Patients With Thumb Carpometacarpal Joint Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Michael Chu Kay MAK, Associate Consultant and Clinical Assistant Professor (Honorary), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT CMCJOA_Protocol_v1
Record Dates: First submitted 2019-12-04; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis Thumb

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor and biostatistician will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arthroscopic Debridement (Active Comparator): Patients who are randomized into this arm will receive arthroscopic debridement
  Interventions: Procedure: Arthroscopic Debridement
- Arthroscopic Hemi-Trapeziectomy with Mini TightRope (Active Comparator): Patients who are randomized into this arm will receive arthroscopic hemi-trapeziectomy with mini tightrope
  Interventions: Procedure: Arthroscopic Hemi-Trapeziectomy with Mini TightRope

INTERVENTIONS:
Procedure: Arthroscopic Debridement — Arthroscopic debridement will be performed under portal site local anaesthesia.
  Arms: Arthroscopic Debridement
Procedure: Arthroscopic Hemi-Trapeziectomy with Mini TightRope — Anaesthesia, position and arthroscopy will be performed in the same way as for arthroscopic debridement, except the distal part of the trapezium will be resected to a depth of 3-4mm together with protruding osteophytes.
  Arms: Arthroscopic Hemi-Trapeziectomy with Mini TightRope

SUMMARY:
Patients with thumb carpometacarpal joint osteoarthritis usually suffer from pain, joint enlargement, inflammation, deformity and loss of function. Conservative treatments usually are the first-line interventions, unfortunately some of the patients do not response to such treatments and surgical treatment will then be considered.

Compare to other traditional surgical techniques, arthroscopic techniques has resulted in the potential to treat osteoarthritis in a minimally invasive approach, avoiding the need for a larger incision. Other advantages of arthroscopy include less scarring and joint contracture, less risk of neurovascular injury, improved appearance, limited morbidity and quicker recovery. Although arthroscopic methods have been proved to be effective, there is lack of high-level evidence based studies to conclude one operation is superior to another. Hence, this study is designed to investigate outcomes of the two arthroscopic surgical methods (arthroscopic debridement vs arthroscopic hemi-trapeziectomy with Mini TightRope). The result of this study is expected to provide significant evidence based clinical data for surgeons worldwide on treating the thumb carpometacarpal joint osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Eaton and Glickel stage II and III of thumb carpometacarpal joint osteoarthritis
* Age≥18 years old
* Failed to response to nonsurgical/conservative treatments including orthoses/splinting, activity modification, oral analgesics (e.g. nonsteroidal anti-inflammatory drugs), strengthening/flexibility exercises, and injections of corticosteroid or hyaluronic acid
* Willing to receive surgery

Exclusion Criteria:

* Patients received previous thumb surgery proximal to the interphalangeal joint (IPJ)
* Patients with prior traumatic thumb injuries (e.g. fracture, dislocation)
* Patients with significant metacarpophalangeal joint (MCPJ) pain
* With concurrent procedures on the thumb, e.g. ganglion removal, trigger thumb release

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) Pain Score at Rest and Exertion | Pre-operative
  Pre-operative VAS pain score at rest and exertion will be measured
Visual Analogue Scale (VAS) Pain Score at Rest and Exertion | Post-op 3 months
  VAS pain score at rest and exertion will be measured post-operatively
Visual Analogue Scale (VAS) Pain Score at Rest and Exertion | Post-op 6 months
  VAS pain score at rest and exertion will be measured post-operatively
Visual Analogue Scale (VAS) Pain Score at Rest and Exertion | Post-op 12 months
  VAS pain score at rest and exertion will be measured post-operatively
Visual Analogue Scale (VAS) Pain Score at Rest and Exertion | Post-op 24 months
  VAS pain score at rest and exertion will be measured post-operatively
Short-Form Survey (SF-36) | Pre-operative
  Generic health status instrument to assess quality of life
Short-Form Survey (SF-36) | Post-op 3 months
  Generic health status instrument to assess quality of life
Short-Form Survey (SF-36) | Post-op 6 months
  Generic health status instrument to assess quality of life
Short-Form Survey (SF-36) | Post-op 12 months
  Generic health status instrument to assess quality of life
Short-Form Survey (SF-36) | Post-op 24 months
  Generic health status instrument to assess quality of life
Disability of Arm, Shoulder and Hand (DASH) questionnaire | Pre-operative
  Specially designed tool to assess upper extremity disability and symptoms
Disability of Arm, Shoulder and Hand (DASH) questionnaire | Post-op 3 months
  Specially designed tool to assess upper extremity disability and symptoms
Disability of Arm, Shoulder and Hand (DASH) questionnaire | Post-op 6 months
  Specially designed tool to assess upper extremity disability and symptoms
Disability of Arm, Shoulder and Hand (DASH) questionnaire | Post-op 12 months
  Specially designed tool to assess upper extremity disability and symptoms
Disability of Arm, Shoulder and Hand (DASH) questionnaire | Post-op 24 months
  Specially designed tool to assess upper extremity disability and symptoms
Patients' Satisfaction Score | Pre-operative
  To grade the subjects' satisfaction regarding to their thumb conditions (0=totally not satisfied; 10=fully satisfied)
Patients' Satisfaction Score | Post-op 3 months
  To grade the subjects' satisfaction regarding to their thumb conditions (0=totally not satisfied; 10=fully satisfied)
Patients' Satisfaction Score | Post-op 6 months
  To grade the subjects' satisfaction regarding to their thumb conditions (0=totally not satisfied; 10=fully satisfied)
Patients' Satisfaction Score | Post-op 12 months
  To grade the subjects' satisfaction regarding to their thumb conditions (0=totally not satisfied; 10=fully satisfied)
Patients' Satisfaction Score | Post-op 24 months
  To grade the subjects' satisfaction regarding to their thumb conditions (0=totally not satisfied; 10=fully satisfied)
Grip Strength | Pre-operative
  Will be measured in kg
Grip Strength | Post-op 3 months
  Will be measured in kg
Grip Strength | Post-op 6 months
  Will be measured in kg
Grip Strength | Post-op 12 months
  Will be measured in kg
Grip Strength | Post-op 24 months
  Will be measured in kg
Key and Tip Pinch | Pre-operative
  Will be measured in kg
Key and Tip Pinch | Post-op 3 months
  Will be measured in kg
Key and Tip Pinch | Post-op 6 months
  Will be measured in kg
Key and Tip Pinch | Post-op 12 months
  Will be measured in kg
Key and Tip Pinch | Post-op 24 months
  Will be measured in kg
Range of Motion (ROM) | Pre-operative
  ROM of interphalangeal joint and metacarpal joint of thumb will be measured
Range of Motion (ROM) | Post-op 3 months
  ROM of interphalangeal joint and metacarpal joint of thumb will be measured
Range of Motion (ROM) | Post-op 6 months
  ROM of interphalangeal joint and metacarpal joint of thumb will be measured
Range of Motion (ROM) | Post-op 12 months
  ROM of interphalangeal joint and metacarpal joint of thumb will be measured
Range of Motion (ROM) | Post-op 24 months
  ROM of interphalangeal joint and metacarpal joint of thumb will be measured
Kapandji Score | Pre-operative
  A tool for assessing the opposition of the thumb
Kapandji Score | Post-op 3 months
  A tool for assessing the opposition of the thumb
Kapandji Score | Post-op 6 months
  A tool for assessing the opposition of the thumb
Kapandji Score | Post-op 12 months
  A tool for assessing the opposition of the thumb
Kapandji Score | Post-op 24 months
  A tool for assessing the opposition of the thumb
Complications | Post-operative up to 2 years
  Any complications related to the surgery will be documented

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No